CLINICAL TRIAL: NCT05500274
Title: Social Network Diffusion of COVID-19 Prevention for Diverse Criminal Legal Involved Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB22-0732; U01MD017414 (NIH)
Record Dates: First submitted 2022-08-05; First posted 2022-08-15 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Educational Status; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Using a two-arm 1:1 randomized controlled trial design, 778 participants were enrolled into either a: 1) COVID-19 prevention education arm (Education Arm) or, 2) a network mobilization change agent intervention (Motivational Arm); the latter is a Type I network intervention that includes specific training on mobilization of network members which we have adapted to COVID-19 from HIV prevention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Arm (Active Comparator): The Education condition will include COVID-19 prevention messaging and an interactive activity reinforcing the messages. Testimonial videos will be played including those that describe the testing experience and motivations for testing. This approach combines self-affirmation with misinformation correction to take advantage of the ability to promote adaptive COVID-19 prevention behaviors.
  Interventions: Other: Education
- Motivational Arm (Active Comparator): Study participants randomized to the Motivational Intervention will receive the intervention using a social network diffusion approach. This is a Type I network intervention that includes specific training on mobilization of network members. The Motivational intervention will be based upon a previous workshop divided into four learning and practice modules.
  Interventions: Other: Motivational

INTERVENTIONS:
Other: Education — Testimonial videos will be played including those that describe the testing experience and their motivations for testing. This approach combines self-affirmation with misinformation correction to take advantage of the ability to promote adaptive COVID-19 prevention behaviors. The self-affirmation activity will always precede the presentation of the testimonial videos as leading with misinformation correction can be construed by some as a threat to one's self-adequacy.
  Arms: Education Arm
Other: Motivational — This is a Type I network intervention that includes specific training on mobilization of network members. Training occurs in a group-based setting of 8-10 enrolled participants facilitated by a community facilitator and Motivational Interviewing trained interventionist. At 30 days, a 15-20-minute phone booster communication session reinforces the intervention content
  Arms: Motivational Arm

SUMMARY:
The "Social network diffusion of COVID-19 prevention for diverse Criminal Legal Involved Communities" study will engage people who have been interacted with law enforcement in COVID-19 prevention (testing and/or vaccination) through social network mobilization combined with theory-driven COVID-19 prevention messaging delivered in an interactive group format. Eligible individuals will be enrolled into a two-arm 1:1 randomized controlled trial design. 800 participants will be enrolled into either a: 1) COVID-19 prevention education arm (Education Arm) or, 2) a network mobilization change agent intervention (Motivational Arm).

DETAILED DESCRIPTION:
The "Social network diffusion of COVID-19 prevention for diverse Criminal Legal Involved Communities" study will implement a situation appropriate COVID-19 testing and vaccination social network diffusion intervention - C3 - building upon RADx-UP Phase I lessons and successful social network prevention interventions developed previously by the research team. C3 Criminal Legal Involved (CLI) populations encompass those non-incarcerated who have experienced recent arrest, incarceration, probation, parole or diversion programs such as drug courts. While increases in COVID-19 testing have been observed among this group, there remain members with limited testing history as well as individuals who are vaccine hesitant. COVID-19 prevention messaging can no longer be simplified to "everyone test and/or everyone vaccinate" as testing and vaccination decisions among community members are sensitive to personal histories (i.e., prior infection), local infection rates (i.e., low rates) and testing/vaccination availability. As COVID-19 prevention efforts have become more complicated (i.e., test if exposed), people tend to focus on the messenger, and particularly those that are close to them. Personal connections and communications within existing personal network structures, such as families, friends and other trusted acquaintances represent the cornerstone to increase situation appropriate testing and overcoming COVID-19 vaccine hesitancy. C3 builds upon RADx-UP I, by using a network diffusion approach facilitated through motivational interviewing purposefully geared to mobilize one's own organic social network to increase context appropriate testing and vaccine uptake. Through this process we will maximize the primary benefit and impact of this type of intervention which also has the intended effect of increasing likelihood that the messenger themselves will undergo the same behavior change that they have been trained to promote. We will leverage infrastructure developed in RADx-UP Phase I, which includes 4 high-impact sites across the Central US from Phase I: Baton Rouge LA, Little Rock AR, Indianapolis IN, and Chicago IL. We will utilize established engagement efforts already in place and continue to fully integrate communities in the strategic application of the intervention. We will use the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework to guide implementation. C3 aims to: Aim 1a. Test the efficacy (3-month situation appropriate testing or vaccination) of a network diffusion intervention (C3) versus an existing COVID-19 testing and vaccine linkage to care intervention among: 1) primary study participants (primary outcome); and 2) secondary study participants connected to primary participants (secondary outcome) using a RCT design. Aim 1b. Explore the mechanisms for differential intervention effects at the individual and network-level that may increase situation appropriate testing and/or vaccination uptake. Aim 2. Examine key RE-AIM components in real time tied to the implementation of the network diffusion intervention (C3).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Spend majority of their time in the metropolitan area or county where recruited
* Primary communication in English
* Previous direct or indirect exposure to law enforcement.

Exclusion Criteria:

* Inability to provide informed consent; and
* Active COVID-19 symptoms per CDC guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 778 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Schneider, MD, Principal Investigator — University of Chicago; Russell Brewer, DrPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1235 participants were screened, 936 were eligible, and 778 consented. Baseline surveys could be completed remotely, but intervention sessions required in-person attendance. Randomization occurred only when participants were physically present. Some participants did not attend due to scheduling conflicts and were not randomized.
Period: Overall Study
Arm/Group | Education Arm | Motivational Arm
Started | 378 | 400
Completed | 295 | 334
Not Completed | 83 | 66
Not completed — Not able to complete the session and follow-up visits. | 7 | 15
Not completed — Lost to Follow-up | 76 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Arm | Motivational Arm | Total
Number analyzed (Participants) | 378 | 400 | 778
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (14.7) | 42.5 (14.5) | 42.9 (14.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 156 | 193 | 349
  Female | 180 | 181 | 361
  Intersex | 0 | 1 | 1
  Unknown, Refused, or Missing | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 67 | 128
  Not Hispanic or Latino | 317 | 333 | 650
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 48 | 61 | 109
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 316 | 334 | 650
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 1 | 11
COVID-19 Testing [Count of Participants; unit: Participants] | 378 | 400 | 778
COVID-19 Vaccination [Count of Participants; unit: Participants] | 378 | 400 | 778

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Testing
Description: Number of participants with at least one test within 3 months of baseline.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Education Arm | Motivational Arm
Number analyzed (Participants) | 378 | 400
Participants | 378 | 400

2. Primary Outcome: COVID-19 Vaccination
Description: Number of participants receiving at least one vaccination within 3 months of baseline.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Education Arm | Motivational Arm
Number analyzed (Participants) | 378 | 400
Participants | 378 | 400

ADVERSE EVENTS:
Time Frame: Each participant will be assessed for adverse events over a specific time period, beginning at their baseline visit. The Time Frame for monitoring adverse events will be up to 12 weeks, which aligns with the study protocol. This period covers the duration from each participant's baseline visit to their final follow-up visit. Adverse events will be systematically monitored through the study completion, which is anticipated to occur by May 31, 2024.
Description: Standard adverse events questionnaire in REDCap
Arm/Group | Education Arm | Motivational Arm
All-Cause Mortality (participants affected / at risk) | 0/378 | 0/400
Serious Adverse Events (participants affected / at risk) | 0/378 | 0/400
Other Adverse Events (participants affected / at risk) | 0/378 | 0/400

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT05500274/Prot_SAP_000.pdf